CLINICAL TRIAL: NCT01178021
Title: Estimating the Risk of Plasmodium Vivax Relapses in Afghanistan
Acronym: VRA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Oxford (Other)
Collaborators: National Malaria and Leishmaniasis Control Program, Afghanistan (Other Government); Mahidol University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BAKMAL0903
Record Dates: First submitted 2010-08-06; First posted 2010-08-09 (Estimated); Last update posted 2019-01-15 (Actual); Status verified 2019-01

CONDITIONS: Vivax Malaria
Keywords: malaria; vivax; relapse
MeSH Terms: conditions — Malaria, Vivax; Malaria; Recurrence | interventions — Chloroquine; Primaquine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Chloroquine (Active Comparator): Standard arm
  Interventions: Drug: Chloroquine
- Chloroquine/Primaquine (Experimental): Chloroquine combined with primaquine
  Interventions: Drug: Chloroquine/Primaquine

INTERVENTIONS:
Drug: Chloroquine — Chloroquine 10 mg/kg on day 0 & 1 and 5mg/kg on day 2
  Arms: Chloroquine
Drug: Chloroquine/Primaquine — Chloroquine 10 mg/kg on day 0 & 1 and 5mg/kg on day 2 Primaquine (if given) 0.25mg/kg/day for 14 days
  Arms: Chloroquine/Primaquine

SUMMARY:
This is an open label two-arm randomized prospective study of two treatments for P. vivax malaria. Patients meeting study inclusion criteria will be enrolled and allocated either chloroquine alone or chloroquine plus primaquine (0.25mg/kg/day for 14 days). Patients will be followed-up for 1 year, with clinical and laboratory examinations at each visit. Patients with recurrent P. vivax infection will be treated with the same medication as initially randomized unless contraindicated. Recurrences in the two arms will be compared to estimate the risk of and mean duration to relapse, classify the relapse pattern as early or late relapse and to estimate the efficacy and safety of the study drugs.

Polymerase Chain Reaction (PCR) analysis will be used as far as possible help to distinguish between relapse and re-infection. Samples for chloroquine pharmacokinetic analysis will be collected on day 7 from each study subject as well as on the day of recurrence if within 8 weeks of chloroquine

DETAILED DESCRIPTION:
Globally more than 100 countries are endemic of malaria and about 60% of world population are at risk of getting the infection while around 10% are harboring malaria parasite in their blood stream. Of the four species of plasmodium that infect humans, Plasmodium vivax is responsible for 50% of all malaria cases outside Africa, and is endemic in the Middle East, Asia and Western Pacific, with a lower prevalence in Central and South America a common cause of malaria in many tropical and subtropical regions. Conventional control methods are rather inefficient for preventing transmission of this species of malaria. This is partly due to the persistence of the infectious reservoir, which take the form of latent hypnozoites in the liver, producing recurrent relapses and opportunities for new transmission for several years after initial infection.

Primaquine (PQ) is the only available drug regimen which can eliminate the persisting liver stages (hypnozoites) of P. vivax,but its use for 14 days is ineffective to prevent relapses at 15 mg daily dose (0.25mg/kg) in Southeast Asia and in Brazil, and at a higher dose of 22.5 mg daily in the Southwest Pacific. Due to high relapse rates, a primaquine regimen of 30 mg daily (0.5 mg/kg) for 14 d is now widely recommended for glucose-6-phosphate dehydrogenase (G6PD) normal patients.

P.vivax is the predominant species in Pakistan and eastern Afghanistan. In this area G6PD deficiency is a common trait (7% in Pakistani and 14% in Afghan Pashtoon respectively). However facilities to test for G6PD deficiency are not available and hence routine administration of primaquine is not recommended in national guidelines because of the risk of severe haemolysis in those who cannot be tested.

Several national malaria programmes in Asia have adopted a truncated 5-day course of PQ for vivax malaria to reduce the risk of haemolysis to reasonable levels and to increases compliance rates. Recently this has been documented as being ineffective at reducing relapse rates amongst Afghan refugees in Pakistan while a supervised 14 day course can significantly reduce the frequency of second and third episodes of disease. This is also confirmed by a study in India. Use of the 14 day course is only recommended where the G6PD status of the individual is known, and, currently, where compliance with the full course can be assured. However supervision of patients for 14 day post presentation is seldom feasible in the majority of settings where vivax malaria predominates. Therefore the supposition that patients in a low literacy population will not comply with a 14 day course of treatment in the absence of supervision needs to be confirmed under normal operational conditions. Compliance in taking the drug cannot be monitored by direct observation or by chemical assay of residues in the blood because such interference may, in itself, affect compliance.

ELIGIBILITY:
Inclusion Criteria:

* Adults and children >6 months
* Negative pregnancy test in women at risk of pregnancy
* Microscopic diagnosis of Plasmodium vivax mono-infection (>200/µl asexual forms)
* Axillary temperature ≥37.5°C or oral/rectal temperature ≥38°C or history of fever within the last 24 hours
* Ability to swallow oral medication
* Participant (or parent/guardian if <18 years old) is willing and able to give written informed consent
* Ability (in the investigator's opinion) and willingness of patient or parent/guardian to comply with all study requirements

Exclusion Criteria:

* Severe malaria (see WHO definition)
* Patients with microscopic diagnosis of co-infection with Plasmodium falciparum
* Haemoglobin concentration <8g/dl
* Presence of any condition which in the judgement of the investigator would place the subject at undue risk or interfere with the results of the study e.g. other acute febrile conditions or chronic disease
* Pregnancy or lactation
* History or phenotypic test compatible with severe G6PD deficiency
* History of hypersensitivity to any of the drugs being tested

Min Age: 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 593 (Actual)
Dates: Start 2009-08 (Actual); Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Secondary vivax attack | 1 year
  Completion of the 1-year (± 1 month) follow-up period without secondary vivax attack

SECONDARY OUTCOMES:
secondary vivax attack | 6 months
  Completion of 6-months (± 1 month) follow-up without secondary vivax attack
G6PD prevalence | Time of enrollment
  G6PD status of patients
Recurrence | 1 year
  Time to first recurrence, median time between episodes of vivax infections and total number of episodes in the follow up period
Days of illness, haematocrit | 1 year
  Overall number of days of illness and haematocrit below 30%
Chloroquine levels | Day 7
  Whole blood chloroquine level at day 7 and any day of recurrence of Plasmodium vivax malaria
Adverse events | 1 year
  Adverse event profiles of chloroquine and primaquine

CONTACTS AND LOCATIONS:
Overall Officials: Ghulam Rahim Awab, MD, Principal Investigator — Mahidol Oxford Tropical Medicine Research Unit
Locations (3):
- Afghanistan (3):
  - Provincial Malaria Control Centers (MRC), Maymana, Faryab Province
  - Provincial Malaria Control Centers (MRC), Jalalabad
  - Provincial Malaria Control Centers (MRC), Kunduz